CLINICAL TRIAL: NCT06445127
Title: Evaluation of Patients With Lupus Nephritis Using Kidney MRI (Magnetic Resonance Imaging)
Status: Terminated | Type: Observational
Why Stopped: Occurrence of unforeseen study issues and a presence of unanticipated risks that cannot be adequately quantified.
Sponsor: Johns Hopkins University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00354110
Record Dates: First submitted 2024-05-13; First posted 2024-06-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Known Lupus Nephritis, with elevated UPCR result: Patients will have one scan at baseline, and one every 4 weeks thereafter for 3 visits. The final imaging session is after 6 months of routine therapy.
- No known lupus nephritis: Patients will have one MRI
- Known Lupus Nephritis, with normal Urine Protein Creatinine Ratio (UPCR) result: Patients will have one scan at baseline, and one every 4 weeks thereafter for 3 visits.

SUMMARY:
This study is being done to find out if a non-invasive Magnetic Resonance Imaging (MRI) examination of the kidneys may be helpful in patients with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults over the age of 18 who have been diagnosed with SLE and are able to undergo a kidney MRI.

Exclusion Criteria:

* Any patient that has undergone a renal transplant.
* Any patient that is receiving renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialty clinic
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Presence of inflammation | Six months
  The presence of inflammation within both kidneys will be measured using MRI.
Presence of fibrosis | Six months
  The presence of fibrosis within both kidneys will be measured using MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Homa Timlin, MD, MSc, MRCP, CCST, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No